CLINICAL TRIAL: NCT05532215
Title: Comparison Between Adjunctive Sublingual Misoprostol Versus Adjunctive Placebo in the Reduction of Intraoperative Blood Loss During Caesarean Section
Brief Title: Sublingual Misoprostol in Reduction of Caesarean Blood Loss
Acronym: SUMIROCBLOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: OZORI EBIOGBO STANLEY (Other Government)
Responsible Party: Sponsor-Investigator, OZORI EBIOGBO STANLEY, DR, Federal Medical Centre, Yenagoa
Organization: Federal Medical Centre, Yenagoa (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMCY/O&G/SUMIROCBLOL/2022
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A hospital's pharmacist/pharmacologist will manufacture the misoprostol tablets at doses of 200 mcg each as well as the placebo tablets (which will contain vitamin B complex excipient only). The misoprostol tablets and placebo tablets will be indistinguishable. Envelopes will be pre-packed, sealed and outwardly labelled by a hospital's pharmacist/pharmacologist who will take no further part in the study.
  Each pre-packed envelope will contain three 200 mcg misoprostol tablets for the misoprostol arm or three placebo tablets (which will contain vitamin B complex excipient only) for the placebo arm.
  The randomization list will be in the possession of a research assistant who will take no further part in the study after randomly allocating the participants to the study arms, till the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol (Experimental): 400 mcg of sublingual misoprostol as two 200 mcg misoprostol tablets at the point of starting the uterine incision at caesarean section, then bolus administration of 10 IU of intravenous oxytocin followed by an infusion of 20 IU of oxytocin in 500 ml of normal saline at a rate of twenty drops per minute to run over eight hours.
  Interventions: Drug: Misoprostol; Drug: Oxytocin
- Placebo (Placebo Comparator): Two sublingual placebo tablets similar to the misoprostol tablets at the point of starting the uterine incision at caesarean section, then bolus administration of 10 IU of intravenous oxytocin followed by an infusion of 20 IU of oxytocin in 500 ml of normal saline at a rate of twenty drops per minute to run over eight hours.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — The misoprostol tablets to be used in the study will be of the same brand and batch
  Arms: Misoprostol
Drug: Oxytocin — The oxytocin ampoules to be used in the study will be of the same brand and batch

SUMMARY:
Caesarean delivery is inevitably associated with a higher amount of blood loss vis-à-vis primary postpartum haemorrhage, when compared to vaginal delivery. Oxytocin use in tropical developing countries for the reduction blood loss at caesarean section have been met with challenges of ineffectiveness due to poor transportation, inadequate storage and drug adulteration. Therefore, there is a need for an effective, temperature stable uterotonic with a lesser risk of adulteration. The study is aimed at evaluating the effectiveness and safety of adjunctive sublingual misoprostol in reducing intraoperative blood loss at caesarean section.

DETAILED DESCRIPTION:
It would be a double blind randomized controlled trial. One hundred and fifty-two pregnant women at term who have indications for caesarean section and have risk factors for primary postpartum haemorrhage, as well as meet the eligibility criteria would be randomized equally into two study arms (Misoprostol study arm and Placebo study arm) after informed consent. The Misoprostol study arm will receive 400 mcg of sublingual misoprostol as two 200 mcg misoprostol tablets. The Placebo study arm would receive two sublingual placebo tablets similar to the misoprostol tablets. The Misoprostol and the Placebo tablets will be given in each study arm at the point of starting the uterine incision at caesarean section. Both study arms would receive routine intravenous oxytocin at the time of clamping of the umbilical cord. The outcome measures will be estimated intraoperative blood loss, the need for additional intraoperative oxytocic, blood transfusion, the occurrence of side effects, and incidence of primary postpartum haemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at term (37+0 weeks to 41+6 weeks gestational age) for elective or non-elective caesarean sections
* Pregnant women who have risk factor for primary postpartum haemorrhage
* Pregnant women who consent to participate in the study

Exclusion Criteria:

* Pregnant women who withhold consent to participate in the study
* Caesarean sections for dire emergencies (umbilical cord prolapse, suspected fetal distress and active antepartum haemorrhage)
* Previous caesarean sections or other uterine surgeries
* Pregnant women with no risk factor for primary postpartum haemorrhage
* Allergy to misoprostol use
* Known history of hepatic, renal and haematological disorders
* Caesarean section to be done under general anaesthesia
* Fever (temperature ≥ 37.5 degrees centigrade)
* Pre-operative anaemia (pre-operative haematocrit level < 30 %)
* Pregnant women who are unconscious or have eclampsia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-10-14 (Estimated); Study Completion 2023-11-14 (Estimated)

PRIMARY OUTCOMES:
Estimated volume of intraoperative blood loss | Immediate postoperative period
  Intraoperative blood loss would be estimated by standard volumetric and gravimetric methods using standard calibrated suction bottles for the volumetric method and for the gravimetric method; wet weight of the abdominal mops, delivery mats, theatre drapes, theatre gowns and vaginal swabs will be gotten using the Mettler PB 153 weighing scale after its re-calibration. The total estimated intraoperative blood loss (T) will be measured by calculating the sum total of the weights of the blood soaked abdominal mops, vaginal gauzes, theatre drapes, theatre gowns and delivery mat (S) and subtracting the sum total of the dry weights of the used abdominal mops, vaginal gauzes, theatre drapes, theatre gowns and delivery mat (D) as shown in the equation: T = S - D. It will be assumed that 1 ml of blood weighs approximately 1 g

SECONDARY OUTCOMES:
Additional intraoperative oxytocic | From intraoperative administration of the study intervention till 4 hours postoperative
  Additional intraoperative oxytocic as10 IU oxytocin when there is absence of uterine tone as assessed by the lead surgeon ten minutes after administration of the intervention drug. Intramuscular ergometrine at a dose of 0.5 mg will be used as a second-line additional uterotonic agent where there are no contraindications.
Postoperative blood transfusion | From intraoperative administration of the study intervention till 48 hours postoperative
  Postoperative blood transfusion indicated by occurrence of primary postpartum haemorrhage (an intraoperative blood loss ≥ 1,000 ml following caesarean section or symptomatic postoperative haematocrit level ≤ 24 %)
Side effect profile | From intraoperative administration of the study intervention till 4 hours postoperative
  Side effect including nausea, vomiting, fever, and shivering
Postoperative haematocrit level | At 48 hours postoperative
  48 hours postoperative haematocrit level

CONTACTS AND LOCATIONS:
Overall Officials: Stanley E Ozori, Principal Investigator — Department of Obstetrics and Gynaecology, Federal Medical Centre, Yenagoa
Locations (1):
- Federal Medical Centre Yenagoa, Yenagoa, Bayelsa State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF